CLINICAL TRIAL: NCT00585897
Title: Title: Effects of Discontinuation of Sugar Sweetened Beverages on Hemoglobin A1c, Fasting and Post Prandial Blood Glucose in Type 2 Diabetics
Brief Title: Effect of Discontinuation of Sugar Sweetened Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00010382
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral counseling (Experimental): Individual sessions which utilize motivational interviewing to assist participants to discontinue sugar sweetened beverages from their diet.
  Interventions: Behavioral: discontinuation of sugar sweetened beverages

INTERVENTIONS:
Behavioral: discontinuation of sugar sweetened beverages — Individual sessions which utilize motivational interviewing to assist participants to eliminate sugar sweetened beverages from their diet.

SUMMARY:
Purpose The purpose of this study is to investigate the effects of discontinuation of sugar sweetened beverages on hemoglobin A1c (HbA1c) and plasma fasting and post-prandial blood glucose in a population with type 2 diabetes.

Hypothesis Elimination of sugar sweetened beverages from the diet for a 4 week period will lead to a decrease in HbA1c and plasma fasting and 2 hour post prandial blood glucose in a population with a history of type 2 diabetes and high consumption of sugar sweetened beverages.

Specific aims to test hypothesis

1. Investigate how elimination of sugar sweetened beverages from the diet affects HbA1c and plasma fasting and two hour post prandial blood glucose.
2. Test the feasibility of carrying out a simple diet intervention in an outpatient population with type 2 diabetes.

DETAILED DESCRIPTION:
Type and Design of Study This will be a pilot study including adult patients age >/= 18 diagnosed with Type 2 Diabetes who are patients at the Duke Outpatient Clinic (DOC) or patients in the general medicine or family practice clinics in Durham County. The intervention will be elimination of sugar sweetened beverages from the diet in a population of type 2 diabetic subjects for four weeks. Sugar sweetened beverages will be defined as any liquid beverage containing calories that can be attributed to natural or added sugar. This will not include beverages that contain mainly artificial sweeteners (e.g.: NutraSweet®, saccharin, Splenda®, or Equal®), plain milk, or water.

ELIGIBILITY:
Inclusion Criteria:

1. Prior diagnosis of Type 2 Diabetes for at least 1 year based on one of the following:

   * Fasting blood glucose >126 on two separate occasions
   * Random blood glucose >200 with symptoms
   * Abnormal 75 or 100 gram Oral Glucose Tolerance Test (OGTT) defined as: fasting blood glucose >100, 2hour post prandial blood sugar of >140
   * On medications for diabetes (oral or insulin)
2. Age >/=18
3. Stable but uncontrolled blood glucose (Hemoglobin A1C >7%, </= 12%)
4. Ingestion of at least three eight ounce servings of sugar sweetened beverage daily.
5. Stable solid diet and exercise pattern and agreement not to change these during the study
6. Able and willing to maintain a complete diet diary for three days each week of the study (total of 12 days of recording)
7. Able to attend regular study visits
8. Able to give informed consent
9. Working phone number in order to contact patient
10. Able and willing to understand and comply with the intervention

Exclusion Criteria:

1. Women who are known to be pregnant at enrollment based on a positive pregnancy test. Pregnancy test will be given to all female subjects of child bearing age prior to enrollment in the study. Pregnant women will be excluded on the basis that blood glucose data are significantly affected by the physiology of pregnancy. This exclusion is not based on any potential risk to the pregnant women or fetus.
2. Individuals <18 years of age
3. Diagnosis of Type 1 Diabetes
4. Malabsorbtive syndrome of any type (will be determined based on medical history from patient and/or medical chart)
5. On Acarbose prior to start of study
6. On a weight loss diet within one month of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 4 weeks for each participant

SECONDARY OUTCOMES:
Fasting glucose | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bryan C. Batch, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Apovian CM. Sugar-sweetened soft drinks, obesity, and type 2 diabetes. JAMA. 2004 Aug 25;292(8):978-9. doi: 10.1001/jama.292.8.978. No abstract available. PMID 15328331
- [Background] Schulze MB, Manson JE, Ludwig DS, Colditz GA, Stampfer MJ, Willett WC, Hu FB. Sugar-sweetened beverages, weight gain, and incidence of type 2 diabetes in young and middle-aged women. JAMA. 2004 Aug 25;292(8):927-34. doi: 10.1001/jama.292.8.927. PMID 15328324